CLINICAL TRIAL: NCT04675580
Title: Tele Toy Talk: Telehealth Language Intervention
Brief Title: Telehealth Language Intervention for Children With Autism Ages 2-4 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-03023432; 19-07020518 (Other: Weill Cornell Medicine IRB)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele Toy Talk (Experimental): Caregivers of child participants receive 1-hour of telemedicine featuring parent-mediated naturalistic developmental behavioral intervention weekly for 10 weeks.
  Interventions: Behavioral: Toy Talk
- Multiple Baseline (No Intervention): Prior to receiving the intervention, participants will be randomized into one of three baseline conditions: a three-, four-, or five-week baseline period. At each weekly baseline session, caregivers will record the Tele-BOSCC (see Outcomes Measures section).

INTERVENTIONS:
Behavioral: Toy Talk — Language modeling strategy encouraging caregivers to (1) talk about the toys the child is playing with, including the states, actions, and properties of the toys and (2) give the object its name using a lexical noun phrase.
  Arms: Tele Toy Talk

SUMMARY:
The main goal of this intervention is to increase caregivers' use of interactive play and communication strategies to improve the child's early sentence development using telemedicine and video-based feedback.

DETAILED DESCRIPTION:
Record was updated 11/2/2021 to include more detailed information about outcome measure time points. Specifically, secondary outcome measures will be collected more frequently over the course of the study (i.e., at baseline [before starting intervention], immediate follow-up [week 12], and long-term follow-up [3 months after intervention] assessments). No changes were made to outcome measures or how they are operationalized.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder (ASD) and/or communication disorder
* Child speaks at least 50 single words or uses emerging word combinations
* Caregivers have Internet availability from their home

Exclusion Criteria:

* Child speaks using complex sentences
* Child is not within 2 to 4 years of age at time of enrollment

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in number of unique combinations of subjects and verbs - caregiver | Baseline (Before starting intervention); Week 4; Week 8; Week 12
  Number of unique combinations of subjects and verbs used by the caregiver at baseline, intervention midpoint, and post-evaluation. This will be calculated by transcribing 12-minute language samples from the BOSCC using Systematic Analysis of Language Transcripts (SALT) software.
Change in number of unique combinations of subjects and verbs - child | Baseline (Before starting intervention); Week 4; Week 8; Week 12
  Number of unique combinations of subjects and verbs used by the child at baseline, intervention midpoint, and post-evaluation. This will be calculated by transcribing 12-minute language samples from the BOSCC using Systematic Analysis of Language Transcripts (SALT) software.
Change in caregiver mean length of utterance | Baseline (before starting intervention); Week 4; Week 8; Week 12
  Mean length of utterance used by caregiver at baseline, intervention midpoint, and post-evaluation. This will be calculated by transcribing 12-minute language samples from the BOSCC using Systematic Analysis of Language Transcripts (SALT) software.
Change in child mean length of utterance | Baseline (before starting intervention); Week 4; Week 8; Week 12
  Mean length of utterance used by child at baseline, intervention midpoint, and post-evaluation. This will be calculated by transcribing 12-minute language samples from the BOSCC using Systematic Analysis of Language Transcripts (SALT) software.
Change in Brief Observation of Social Communication Change (BOSCC) scores | Baseline (before starting intervention); Week 4; Week 8; Week 12
  Child's scores on the Brief Observation of Social Communication Change (BOSCC) at baseline, intervention midpoint, and post-evaluation. BOSCC scores are not linear. Each item is rated on a 6-point scale from 0 (abnormality is not present) to 5 (abnormality is present and significantly impairs functioning).

SECONDARY OUTCOMES:
Change in scores on the Observation of Spontaneous Expressive Language (OSEL) - baseline | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention)
  Child's scores on the Observation of Spontaneous Expressive Language at baseline, post-evaluation, and long-term follow-up evaluation (3 months after ending intervention). Scores on the OSEL are not linear. Scores range from 0 to 3, with higher scores indicating more impairment.
Change in scores on the Vineland-3 | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention)
  Scores on the Vineland-3 at baseline, post-evaluation, and long-term follow-up evaluation (3 months after ending intervention). The Vineland-3 provides norm-referenced scaled scores for 11 skill areas (M = 10; SD = 3) as well as standard scores (M =100, SD = 15) for three adaptive domains.

OTHER OUTCOMES:
Change in scores on the Acceptance and Action Questionnaire, Second Version (AAQ-II) | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention).
  Caregiver scores on the Acceptance and Action Questionnaire, Second Version (AAQ-II) at baseline, post-evaluation, and long-term follow-up evaluation (3 months after end of intervention). Items are rated on a Likert-type scale of 1 through 7, and scores range from 7 to 49.
Change in scores on the Emotion Regulation Questionnaire (ERQ) | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention).
  Caregiver scores on the Emotion Regulation Questionnaire (ERQ) at baseline, post-evaluation, and long-term follow-up evaluation (3 months after ending intervention). The ERQ is a 10-item scale with each item consisting of a 7-point Likert-type scale ranging from 1 to 7.
Change in scores on the Caregiver Strain Questionnaire - Short Form 7 (CSQ-SF 7) | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention).
  Scores on the Caregiver Strain Questionnaire - Short Form 7 (CSQ-SF 7) at baseline, post-evaluation, and long-term follow-up evaluation (3 months after ending intervention). The CSQ-SF7 contains seven items, with response options on a five-point Likert-type scale.
Change in scores on the Parent Stress Index-4th Edition (PSI-4) | Baseline (before starting intervention); Week 12; Follow-up assessment (3 months after end of intervention).
  Scores on the Parent Stress Index (PSI-4) at baseline, post-evaluation, and long-term follow-up evaluation (3 months after ending intervention). The PSI-4 is a 120-item inventory that provides two domain scores that are quantified using T scores (mean of 50; standard deviation of 10).

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Kim, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center for Autism and the Developing Brain/New York-Presbyterian Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No